CLINICAL TRIAL: NCT02313662
Title: Trimodalitets-studie Hvidt Lys vs. NBI vs. PDD Ved Detektion af Flad Dysplasi og CIS Ved TURB
Brief Title: Comparison of White Light, PDD and NBI in Detection of Flat Dysplasia and CIS at TURB - a Study of Trimodality
Acronym: DaBlaCa-8
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Herlev Hospital (Other); Hospitalsenheden Vest (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jørgen Bjerggaard Jensen, Professor, Aarhus University Hospital
Other Study IDs: DaBlaCa-8
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Narrow Band Imaging and PDD in Cystoscopy
MeSH Terms: interventions — Narrow Band Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: NBI and PDD

SUMMARY:
All patients planned for PDD guided TURB can be included in this study. Two different optics with PDD and NBI are applied to the resectoscope in addition to regular WL.

First, a WL cystoscopy is made and any suspect areas are noted on the registration form, then NBI is used and any suspect areas are noted and finally the cystoscopy is made with PDD with registration of any additional findings. To adjust for bias introduced by photo bleaching, the second part of the study will be performed with PDD as the second modality. Any flat lesions will be biopsied if they appear suspicious in one of the modalities.

The registration form is completed by the surgeon, once the pathology results are known.

A total number of 152 patients is planned to be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PDD according to the Danish guidelines

Exclusion Criteria:

* Patients not fulfilling the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PDD according to the Danish guidelines
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Detection of CIS | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Bjerggaard Jensen, Principal Investigator — University of Aarhus
Locations (4):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Herlev
  - Hospitalsenheden Vest, Holstebro
- Oslo University Hospital, Oslo, Norway